CLINICAL TRIAL: NCT05165888
Title: Targeting Bias to Reduce Disparities in End of Life Care: Clinician Communication Behavior in Simulated Patient Encounters Study
Brief Title: Targeting Bias to Reduce Disparities in End of Life Care
Acronym: BRiDgE-Sim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); University of Nebraska Lincoln (Other); Tulane University School of Medicine (Other); Dartmouth College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2021-12898; 5K23MD015277-03 (NIH)
Record Dates: First submitted 2021-11-10; First posted 2021-12-21 (Actual); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Terminal Illness; Critical Illness
Keywords: Palliative; Communication
MeSH Terms: conditions — Critical Illness; Communication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communication and Bias Mitigation Training (Experimental): This is a communication training session based on a culturally-based program developed with rural, southern Black patients and families and modified for an urban, northern population. A strategy of bias mitigation successfully used with medical students will be adapted for practicing clinicians using results of phase 1. This strategy is based on transformational learning theory and incorporates critical reflection, guided dialogue, perspective taking exercises, role plays and strategy development. If specific communication behaviors are found related to bias and stereotyping in phase 1, these will be discussed and targeted using these techniques. Otherwise, these techniques will be used to address racial bias generally. The intervention will be incorporated within the communication training session.
  Interventions: Behavioral: Communication and Bias Mitigation Training
- Communication Training Only (Active Comparator): This is a communication training session based on standard palliative care techniques to listen empathically, share prognostic information and treatment options, elicit patient and family goals and values related to their treatment, and facilitate shared decision-making regarding end-of-life treatment.
  Interventions: Behavioral: Communication skills training

INTERVENTIONS:
Behavioral: Communication and Bias Mitigation Training — Training to improve communication skills and reduce the effect of racial bias on clinician communication behavior
  Arms: Communication and Bias Mitigation Training
Behavioral: Communication skills training — Training to improve communication skills between physicians and caregivers.
  Arms: Communication Training Only

SUMMARY:
This study aims to determine the ways in which clinician implicit racial biases affect clinician communication with family members of patients near the end of life and to test a novel physician training intervention to reduce the effects of implicit racial bias on quality of communication.

Phase 1:

A sample of 50 physicians who care for seriously ill patients, including oncologists, critical care physicians and hospital-based internists will participate in a simulated clinical encounter with a Black standardized family member (actor) of a hypothetical case patient. Measures of implicit and explicit bias will be correlated with verbal and nonverbal communication behavior.

Phase 2:

This is a 2-arm randomized feasibility pilot of an intervention to mitigate the effects of clinician implicit bias on communication behavior. Physicians who treat patients with serious illness including oncologists, critical care physicians and hospital-based internists will be recruited to participate in a communication training session to reduce the effects of implicit bias or a control training session focusing only on communication skills. Their communication behavior will be videotaped during a simulated encounter with a Black standardized family member (actor) of a hypothetical patient with serious illness before and after the training sessions. The communication behavior before and after the training session will be compared between physicians that received the communication skills only intervention versus the physicians that received the communication skills and bias mitigation training.

The primary hypothesis is that physicians who receive both the communication skills and the bias mitigation training will have greater improvements in communication skills with the Black standardized caregiver (actor) compared with those who receive only the communication skills training.

This registration is inclusive of phase 2 only as phase 2 is the clinical trial portion of this research. Phase 1 is not a clinical trial as it was an observational study that did not include an intervention. Phase 1 data was used to inform the structure and analysis of phase 2.

DETAILED DESCRIPTION:
Significance

Scope of the problem:

US adults over 65 are more racially diverse than ever, and this trend will continue. The number of older Black Americans is projected to reach 12 million or 12% of older adults by 2060. Although the growth of palliative care has improved the quality of end-of-life care over the past two decades, racial and ethnic minority patients have not fully benefitted from these advances. There are well-documented disparities in access and uptake of palliative care and in the quality and intensity of end-of-life care. These inequalities affect many minority groups, each with its unique history, language and culture that may influence the underlying mechanisms of disparities. The current proposal focuses on Black Americans who experience disparities that are deeply rooted in complex historical and present-day interactions with the health care system.

Mechanisms underlying disparities in quality of end-of-life care

Clinician factors:

There is a major gap in knowledge regarding clinicians' contributions to end-of-life disparities. Most physicians in the US are White, and only 4% are Black. Patient-physician racial discordance is associated with decreased quality of communication. Clinician communication during racially discordant encounters is an important and modifiable factor in end-of-life care disparities.

End-of-life conversations are less likely to result in goal-concordant care for Black compared with White patients. Possible explanations for these differences include implicit bias as well as explicit beliefs. Stereotypical beliefs hinder development of true knowledge of the patient by shortcutting around knowledge-gathering communication. Implicit attitudes decrease the quality of communication affecting partnership, respect, affiliation and trust. Reduced access to quality communication could explain some of the increased use of aggressive care and reduced quality of end-of-life care for Black patients.

Bias and Communication:

Implicit bias refers to unconscious, automatic positive or negative attitudes. Clinicians rarely mention race and ethnicity as barriers to communication, suggesting that they are unable to name these barriers due either to the implicit nature of the bias or to social desirability bias in reporting. The Implicit Association Test (IAT) demonstrates unconscious racial bias among clinicians. Implicit bias predicts patient ratings in domains critical to quality end-of-life care including interpersonal treatment, communication and trust. Physician implicit bias results in poor communication patterns, and poor patient-doctor relationships. Some physicians express explicit beliefs regarding Black patients' "resistance" to hospice care. It is unknown whether explicit stereotypes about end-of-life preferences influence communication behavior.

Bias Mitigation:

Evidence-based strategies have been developed to reduce effects of implicit bias, but few have been systematically tailored to gaps in care and measured for effectiveness in the clinical setting. There is limited evidence to support specific strategies to reduce the effects of clinician bias on clinical care. Strategies that focus only on making clinicians aware of their biases are unlikely to reduce their effects in the long term without providing them with specific strategies to overcome them. A strategy based on transformative learning theory and incorporating critical reflection, guided dialogue, perspective taking exercises, role plays and strategy development has been successfully used with medical students.

Aims/Objectives:

The aim of this study is to assess the effects of clinician racial bias on end-of-life communication and to develop interventions to reduce the effects of implicit bias on quality of clinician communication. There are two study objectives: (1) Establish which communication behaviors in the end-of-life setting are most affected by clinician implicit racial bias and explicit stereotyping. (2) Pilot a theory-driven intervention to improve clinician communication and reduce disparities in quality end-of-life care. These objectives will be met in two study phases.

Methods/Design:

Phase 1:

Methods:

(1) The investigators will develop a case depicting a hospitalized 72-year-old with lung cancer and sepsis due to pneumonia on high-flow nasal cannula with my mentorship team of experts in palliative medicine and critical care. The investigators will design a clinical encounter with the caregiver to discuss goals of care. 2) The caregiver encounter will be piloted with critical care and hospitalist physicians at Montefiore to ensure realism and achieve standardization. Black standardized caregivers will be recruited from the pool of actors used by the Einstein Clinical Skills Center. (3) Standardized caregivers will be trained in the use of a communication assessment tool. (4) 50 physicians will be recruited to participate in a videotaped high-fidelity simulation of the encounter. The session will be followed by a 1-hour communication skills training. (5) Immediately after the simulation subjects will complete the IAT and a questionnaire probing for attitudes about race and end-of-life care along with demographic questions. The investigators will assess training needs by adapting a previously developed questionnaire measuring physicians' self-identified serious illness communication training needs by incorporating questions about bias mitigation skills. The IAT is publicly available here: https://implicit.harvard.edu/implicit/selectatest.html.

COVID-19 Concerns:

The Clinical Skills Center will be holding in-person simulations with standardized patients for the purposes of medical education starting in May 2021. The simulations in this study will not begin until after that time and will involve less risk than typical simulations because they will not entail a physical examination of the standardized caregiver. Actors and participants will be equipped with personal protective equipment including surgical masks. Trainers and participants in the training session will be required to wear provided surgical masks and remain six feet apart during the training sessions. If COVID-19 state or institutional guidelines prohibit these types of encounters at the time the simulations will be launched, the simulations and training will be adapted to a virtual format and nonverbal behavior coding will be adjusted. These changes will be submitted to the Institutional Review Board (IRB) as an amendment.

Data collection:

Encounters will be videotaped. The amount of time the physician and standardized caregiver speak will be recorded. A five-point verbal communication rating scale will be used to rate physician (1) informativeness, (2) supportiveness, and (3) partnership-building and a modified version of the Nonverbal Accommodation Analysis System (NAAS). The NAAS will be modified to include physical distance and open/closed body language which were shown to be important in serious illness encounters.

Another questionnaire will be administered at the end of the training. The investigators will ask physicians to rate their experiences with different educational modalities presented in the training session, such as feedback from observed encounters, communication drills and role-plays. In addition, the questionnaire will include the cognitive and affective empathy portions of the Interpersonal Reactivity Index. For participants in the active group only, several questions will assess the illusion of ownership of the virtual body in the VR experience. Open-ended questions will be used to gather formative information that the researchers may not have considered. This questionnaire will be distributed at the end of the communication skills training.

Analysis plan:

Bivariate associations of communication scores with IAT scores will be estimated with Pearson or Spearman rank correlation coefficients depending on the distribution of the data. Generalized linear models (GLM) will be fit to the data to assess the associations of the IAT and racial attitudes with primary and secondary communication outcomes, while controlling for potential confounding variables including clinician age, gender and specialty. The identity link will be used in the GLM for continuous communication outcomes. Subgroup analysis will be performed in Asian, Black and Hispanic physicians if there are sufficient numbers in these groups to assess heterogeneity of the associations by race.

Power analysis:

The target sample size of 50 participants would have >80% power to detect a minimum correlation between IAT score and verbal dominance of ρ ≥ 0.38 using a two-sided hypothesis test of a single correlation with a significance level of 0.05. This correlation is similar in magnitude to associations observed in prior studies; B=11.0 in one study and r = 0.32 in another.

Phase 2:

Methods:

This is a communication training session based on a culturally-based program developed with rural, southern Black patients and families and modified for an urban, northern population. A strategy of bias mitigation successfully used with medical students will be adapted for practicing clinicians using results of phase 1. This strategy is based on transformative learning theory and incorporates critical reflection, guided dialogue, perspective taking exercises, role plays and strategy development. In this study, a virtual reality (VR) experience (https://michigan.it.umich.edu/news/2023/07/31/education-andawareness- in-vr-new-experience-illustrates-the-effects-of-racial-discrimination/) will be used as the disorienting dilemma to spark the process of transformative learning. This brief experience embodies the participant in the experiences of an African American man over their life course. It is aimed to engender empathy and perspective taking. Following the VR experience, participants will debrief with the facilitator in small groups, discuss how implicit bias impacts the clinical encounter, brainstorm bias mitigation techniques and role-play strategies to mitigate bias in the clinical encounter. If specific communication behaviors are found related to bias and stereotyping in phase 1, these will be discussed and targeted using these techniques. Otherwise, these techniques will be used to address racial bias generally. The intervention will be incorporated within the communication training session.

Design:

Clinicians will be randomized 1:1 to the active intervention or a control communication training without bias mitigation techniques. Allocation concealment will be in place to ensure the individual enrolling the subject into the study has no a priori knowledge of group assignment. Block randomization will occur with randomly mixed block sizes of 2, 4, and 6. The allocator (research assistant) will hide block size from the executor (PI) in order to prevent the executor from predicting the next assignment. Randomization will be carried out by having a piece of paper that has the phrase "Intervention (Communication + Bias)" or "Control (Communication only)" placed inside an opaque envelope. The outside of the envelopes will be labeled with the sequence number. After a subject has been enrolled into the study and consented, the next sequence numbered envelope on the stack will be opened to determine the study group that the subject will enter.

Participants will be videotaped during high-fidelity simulations of encounters with caregivers described in phase 1, before and after receiving the intervention or control. The intervention and simulations will take place in one half-day workshop.

Study population and Recruitment:

A new group of intensivists, oncologists and hospitalists will be recruited. Physician subjects will be recruited face-to-face by the PI, through departmental email blasts and emails to contacts of the study team. As in phase 1, physicians will complete a screening questionnaire to exclude those that do not routinely encounter hospitalized patients with a life expectancy of less than one year. Potential subjects will be asked about the frequency and timing of previous communication and bias training. Physicians practicing Hospice and Palliative Medicine will be excluded because of their extensive prior training in communication.

Data collection:

Encounters will be videotaped. The investigators will use the five-point verbal communication rating scale and a modified version of the NAAS for nonverbal communication behaviors during the standardized encounter as described in phase 1 above. A research assistant who did not participate in the training sessions and is blinded to participant group will code communication behaviors. Subjects will complete the IAT and the questionnaire described in phase 1 immediately after the first encounter.

Analysis plan:

Initially, the mean change in verbal and nonverbal communication scores pre- and post-intervention will be evaluated within each intervention arm using paired t-tests or Wilcoxon tests if the data are not normally distributed. To assess whether communication scores improved more in the bias mitigation treatment compared with communication training only control, a generalized linear model will be fit to the data with post-intervention score as the outcome, and pre-intervention score and intervention arm as the main effects. In addition, the investigators will explore whether pre-intervention level of bias modifies the effect of bias mitigation training, e.g., those with more bias will have a greater difference in improvement between the intervention and control group, by including in the model an interaction term between IAT score and treatment group on communication scores. A positive interaction will indicate that implicit bias as measured by the IAT modifies the effect of treatment group on communication score. With 25 subjects per intervention arm, the study will have 80% power to detect an effect size of 0.8 between groups in pre-post change in communication scores with a two-sided Type 1 error rate of 5%. While this is considered a large effect size according to Cohen's criteria, this is a pilot study in which the primary goal is to assess feasibility and to generate preliminary data on the effect of the proposed communication training intervention for clinicians to mitigate the effects of implicit bias.

Data Management/Analysis:

Communication behavior codes and data from the questionnaires and IAT stored on Montefiore's secure Box drive and will only be accessible by members of the research team. Video recordings will be stored on a password-protected hard drive accessible only to the research team.

Risks/Benefits:

Potential risks: This research poses two main risks to subjects: 1) emotional distress and 2) risk to privacy. There may be some emotional distress caused by learning about one's unconscious racial biases. Emotional distress may also result from passive deception; subjects will not be told that racial bias is the focus of the study until after the intervention. Privacy risk arises because racial biases may be considered sensitive information about the subject.

Adequacy of Protection Against Risks Recruitment and Informed Consent: All subjects will be recruited by the PI through departmental email blasts, emails to contacts of the study team and departmental faculty meeting presentations. The consent process will take place in the Clinical Skills Center on the prior to the standardized patient encounter. Subjects will be informed of their right to participate or discontinue participation at any time without jeopardizing their employment, professional position or relationships with colleagues. Copies of the signed consent form will be given to the subject and placed in the subject's research folder in a locked file drawer in an office in the PI's office expressly designed for this purpose.

Incomplete disclosure of information during the consenting process: Subjects will be informed that they are participating in a study exploring physician cognition, cognitive biases and communication behavior. They will be informed that study participation includes completion of an on-line instrument after the standardized patient encounter. They will not be told during the consent process that implicit racial bias and stereotyping are the focus of the study.

Protections against risks: Personal identifiers not be collected in the on-line instrument; instead a unique study ID will be assigned to each participant. Video recordings will be maintained in a password protected digital folder on a hard drive in a locked office. This database of coded communication scores will be stripped of participant identifiers as soon as all data is collected, and a file linking the study ID and patient identifiers will be kept in a separate, password protected digital folder.

Debriefing: After completion of the on-line bias measurement instrument, the subjects will be shown a debriefing statement including full disclosure of the aims of the study and the intent to examine the relationship between implicit racial bias and stereotyping and communication behavior. This statement will include a reminder that they may discontinue participation at any time and request that their data be removed from the dataset without penalty. The PIs contact information will be provided.

Potential Benefits of the Proposed Research: Subjects are not expected to directly benefit from this research. Importance of the knowledge to be gained: The information from this study will provide knowledge about the role of implicit bias and stereotyping in communication behaviors that have profound effects on the quality of end-of-life care for Black patients. It will also inform efforts to mitigate the effects of this bias in future studies.

Necessity of withholding information in the consent process: Withholding of complete information from the consent process is only acceptable if there is no reasonably effective alternative to achieve the goals of the research. In this case, knowledge of the intent to study implicit racial bias is likely to affect the way physicians communicate in the standardized patient encounter, thus invalidating the results of the study.

ELIGIBILITY:
Inclusion Criteria:

* Practicing physicians
* Specializes in oncology, critical care, hospitalist medicine, emergency medicine or geriatrics

Exclusion Criteria:

* Physicians who do not care for seriously ill patients in the hospital at least 10% of their working time.
* Physicians trained in Hospice and Palliative Medicine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Chuang, MD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Montefiore Medical Center is an institutional member and Dr. Chuang is an individual member of the Palliative Care Research Cooperative (PCRC). The PCRC is funded by the National Institute of Nursing Research (NINR) and is committed to assisting investigators in complying with data sharing policies. The PCRC collects and houses de-identified qualitative and quantitative data from completed research projects. These data are housed within the PCRC Data Repositories. Researchers may access this data consistent with IRB/CHR rules, local, state, and Federal laws and regulations, and the HIPAA Privacy Rule. Investigators may request access to the de-identified PCRC Data Repositories for secondary data analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available at the completion of data analysis and dissemination for the studies, within two years of study completion and will remain available indefinitely.
Access Criteria: Investigators must submit their analysis proposal to the PCRC which will review the request for scientific integrity, feasibility, and analytic rigor and IRB approval or exempt status.

REFERENCES:
- [Background] Lee JJ, Long AC, Curtis JR, Engelberg RA. The Influence of Race/Ethnicity and Education on Family Ratings of the Quality of Dying in the ICU. J Pain Symptom Manage. 2016 Jan;51(1):9-16. doi: 10.1016/j.jpainsymman.2015.08.008. Epub 2015 Sep 16. PMID 26384556
- [Background] Johnson KS. Racial and ethnic disparities in palliative care. J Palliat Med. 2013 Nov;16(11):1329-34. doi: 10.1089/jpm.2013.9468. Epub 2013 Sep 27. PMID 24073685
- [Background] Welch LC, Teno JM, Mor V. End-of-life care in black and white: race matters for medical care of dying patients and their families. J Am Geriatr Soc. 2005 Jul;53(7):1145-53. doi: 10.1111/j.1532-5415.2005.53357.x. PMID 16108932
- [Background] Byrd WM, Clayton LA. Race, medicine, and health care in the United States: a historical survey. J Natl Med Assoc. 2001 Mar;93(3 Suppl):11S-34S. PMID 12653395
- [Background] Feagin J, Bennefield Z. Systemic racism and U.S. health care. Soc Sci Med. 2014 Feb;103:7-14. doi: 10.1016/j.socscimed.2013.09.006. PMID 24507906
- [Background] Connor SR, Elwert F, Spence C, Christakis NA. Racial disparity in hospice use in the United States in 2002. Palliat Med. 2008 Apr;22(3):205-13. doi: 10.1177/0269216308089305. PMID 18477714
- [Background] Smith-Howell ER, Hickman SE, Meghani SH, Perkins SM, Rawl SM. End-of-Life Decision Making and Communication of Bereaved Family Members of African Americans with Serious Illness. J Palliat Med. 2016 Feb;19(2):174-82. doi: 10.1089/jpm.2015.0314. PMID 26840853
- [Background] Kwak J, Haley WE. Current research findings on end-of-life decision making among racially or ethnically diverse groups. Gerontologist. 2005 Oct;45(5):634-41. doi: 10.1093/geront/45.5.634. PMID 16199398
- [Background] Allen RS, Allen JY, Hilgeman MM, DeCoster J. End-of-life decision-making, decisional conflict, and enhanced information: race effects. J Am Geriatr Soc. 2008 Oct;56(10):1904-9. doi: 10.1111/j.1532-5415.2008.01929.x. Epub 2008 Sep 4. PMID 18775035
- [Background] Benton K, Stephens J, Vogel R, Ledlow G, Ackermann R, Babcock C, McCook G. The influence of race on end-of-life choices following a counselor-based palliative consultation. Am J Hosp Palliat Care. 2015 Feb;32(1):84-9. doi: 10.1177/1049909113506782. Epub 2013 Oct 1. PMID 24085311
- [Background] Mack JW, Paulk ME, Viswanath K, Prigerson HG. Racial disparities in the outcomes of communication on medical care received near death. Arch Intern Med. 2010 Sep 27;170(17):1533-40. doi: 10.1001/archinternmed.2010.322. PMID 20876403
- [Background] Sanders JJ, Johnson KS, Cannady K, Paladino J, Ford DW, Block SD, Sterba KR. From Barriers to Assets: Rethinking factors impacting advance care planning for African Americans. Palliat Support Care. 2019 Jun;17(3):306-313. doi: 10.1017/S147895151800038X. Epub 2018 Jun 5. PMID 29869594
- [Background] Mack JW, Weeks JC, Wright AA, Block SD, Prigerson HG. End-of-life discussions, goal attainment, and distress at the end of life: predictors and outcomes of receipt of care consistent with preferences. J Clin Oncol. 2010 Mar 1;28(7):1203-8. doi: 10.1200/JCO.2009.25.4672. Epub 2010 Feb 1. PMID 20124172
- [Background] Cooper LA, Roter DL, Johnson RL, Ford DE, Steinwachs DM, Powe NR. Patient-centered communication, ratings of care, and concordance of patient and physician race. Ann Intern Med. 2003 Dec 2;139(11):907-15. doi: 10.7326/0003-4819-139-11-200312020-00009. PMID 14644893
- [Background] Barnato AE. Challenges In Understanding And Respecting Patients' Preferences. Health Aff (Millwood). 2017 Jul 1;36(7):1252-1257. doi: 10.1377/hlthaff.2017.0177. PMID 28679812
- [Background] Wagner GJ, Riopelle D, Steckart J, Lorenz KA, Rosenfeld KE. Provider communication and patient understanding of life-limiting illness and their relationship to patient communication of treatment preferences. J Pain Symptom Manage. 2010 Mar;39(3):527-34. doi: 10.1016/j.jpainsymman.2009.07.012. Epub 2010 Feb 19. PMID 20171827
- [Background] Gramling R, Gajary-Coots E, Cimino J, Fiscella K, Epstein R, Ladwig S, Anderson W, Alexander SC, Han PK, Gramling D, Norton SA. Palliative Care Clinician Overestimation of Survival in Advanced Cancer: Disparities and Association With End-of-Life Care. J Pain Symptom Manage. 2019 Feb;57(2):233-240. doi: 10.1016/j.jpainsymman.2018.10.510. Epub 2018 Nov 1. PMID 30391655
- [Background] Ingersoll LT, Alexander SC, Priest J, Ladwig S, Anderson W, Fiscella K, Epstein RM, Norton SA, Gramling R. Racial/ethnic differences in prognosis communication during initial inpatient palliative care consultations among people with advanced cancer. Patient Educ Couns. 2019 Jun;102(6):1098-1103. doi: 10.1016/j.pec.2019.01.002. Epub 2019 Jan 2. PMID 30642715
- [Background] Rhodes RL, Batchelor K, Lee SC, Halm EA. Barriers to end-of-life care for African Americans from the providers' perspective: opportunity for intervention development. Am J Hosp Palliat Care. 2015 Mar;32(2):137-43. doi: 10.1177/1049909113507127. Epub 2013 Oct 4. PMID 24097838
- [Background] Cicolello K, Anandarajah G. Multiple Stakeholders' Perspectives Regarding Barriers to Hospice Enrollment in Diverse Patient Populations: A Qualitative Study. J Pain Symptom Manage. 2019 May;57(5):869-879. doi: 10.1016/j.jpainsymman.2019.02.012. Epub 2019 Feb 18. PMID 30790720
- [Background] Barnato AE, Mohan D, Downs J, Bryce CL, Angus DC, Arnold RM. A randomized trial of the effect of patient race on physicians' intensive care unit and life-sustaining treatment decisions for an acutely unstable elder with end-stage cancer. Crit Care Med. 2011 Jul;39(7):1663-9. doi: 10.1097/CCM.0b013e3182186e98. PMID 21460710
- [Background] Chuang E, Hope AA, Allyn K, Szalkiewicz E, Gary B, Gong MN. Gaps in Provision of Primary and Specialty Palliative Care in the Acute Care Setting by Race and Ethnicity. J Pain Symptom Manage. 2017 Nov;54(5):645-653.e1. doi: 10.1016/j.jpainsymman.2017.05.001. Epub 2017 Jul 29. PMID 28760524
- [Background] Elliott AM, Alexander SC, Mescher CA, Mohan D, Barnato AE. Differences in Physicians' Verbal and Nonverbal Communication With Black and White Patients at the End of Life. J Pain Symptom Manage. 2016 Jan;51(1):1-8. doi: 10.1016/j.jpainsymman.2015.07.008. Epub 2015 Aug 20. PMID 26297851
- [Background] Maina IW, Belton TD, Ginzberg S, Singh A, Johnson TJ. A decade of studying implicit racial/ethnic bias in healthcare providers using the implicit association test. Soc Sci Med. 2018 Feb;199:219-229. doi: 10.1016/j.socscimed.2017.05.009. Epub 2017 May 4. PMID 28532892
- [Background] Sabin J, Nosek BA, Greenwald A, Rivara FP. Physicians' implicit and explicit attitudes about race by MD race, ethnicity, and gender. J Health Care Poor Underserved. 2009 Aug;20(3):896-913. doi: 10.1353/hpu.0.0185. PMID 19648715
- [Background] Penner LA, Dovidio JF, Gonzalez R, Albrecht TL, Chapman R, Foster T, Harper FW, Hagiwara N, Hamel LM, Shields AF, Gadgeel S, Simon MS, Griggs JJ, Eggly S. The Effects of Oncologist Implicit Racial Bias in Racially Discordant Oncology Interactions. J Clin Oncol. 2016 Aug 20;34(24):2874-80. doi: 10.1200/JCO.2015.66.3658. Epub 2016 Jun 20. PMID 27325865
- [Background] FitzGerald C, Hurst S. Implicit bias in healthcare professionals: a systematic review. BMC Med Ethics. 2017 Mar 1;18(1):19. doi: 10.1186/s12910-017-0179-8. PMID 28249596
- [Background] Johnson RL, Roter D, Powe NR, Cooper LA. Patient race/ethnicity and quality of patient-physician communication during medical visits. Am J Public Health. 2004 Dec;94(12):2084-90. doi: 10.2105/ajph.94.12.2084. PMID 15569958
- [Background] Cooper LA, Roter DL, Carson KA, Beach MC, Sabin JA, Greenwald AG, Inui TS. The associations of clinicians' implicit attitudes about race with medical visit communication and patient ratings of interpersonal care. Am J Public Health. 2012 May;102(5):979-87. doi: 10.2105/AJPH.2011.300558. Epub 2012 Mar 15. PMID 22420787
- [Background] Blair IV, Steiner JF, Fairclough DL, Hanratty R, Price DW, Hirsh HK, Wright LA, Bronsert M, Karimkhani E, Magid DJ, Havranek EP. Clinicians' implicit ethnic/racial bias and perceptions of care among Black and Latino patients. Ann Fam Med. 2013 Jan-Feb;11(1):43-52. doi: 10.1370/afm.1442. PMID 23319505
- [Background] Teal CR, Gill AC, Green AR, Crandall S. Helping medical learners recognise and manage unconscious bias toward certain patient groups. Med Educ. 2012 Jan;46(1):80-8. doi: 10.1111/j.1365-2923.2011.04101.x. PMID 22150199
- [Background] Gonzalez CM, Kim MY, Marantz PR. Implicit bias and its relation to health disparities: a teaching program and survey of medical students. Teach Learn Med. 2014;26(1):64-71. doi: 10.1080/10401334.2013.857341. PMID 24405348
- [Background] Gonzalez CM, Walker SA, Rodriguez N, Karp E, Marantz PR. It Can Be Done! A Skills-Based Elective in Implicit Bias Recognition and Management for Preclinical Medical Students. Acad Med. 2020 Dec;95(12S Addressing Harmful Bias and Eliminating Discrimination in Health Professions Learning Environments):S150-S155. doi: 10.1097/ACM.0000000000003697. PMID 32889927
- [Background] D'Agostino TA, Bylund CL. Nonverbal accommodation in health care communication. Health Commun. 2014;29(6):563-73. doi: 10.1080/10410236.2013.783773. Epub 2013 Oct 18. PMID 24138223
- [Background] Elk R, Emanuel L, Hauser J, Bakitas M, Levkoff S. Developing and Testing the Feasibility of a Culturally Based Tele-Palliative Care Consult Based on the Cultural Values and Preferences of Southern, Rural African American and White Community Members: A Program by and for the Community. Health Equity. 2020 Mar 26;4(1):52-83. doi: 10.1089/heq.2019.0120. eCollection 2020. PMID 32258958
- See also: Diversity in the Physician Workforce: Facts & FIgures 2014. American Association of Medical Colleges — https://www.aamc.org/data-reports/workforce/report/diversity-facts-figures

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Communication and Bias Mitigation Training | Communication Training Only
Started | 11 | 11
Completed | 11 | 10 (One subject did not complete the post-intervention measures because they had to leave the lab early due to a scheduling conflict.)
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Communication and Bias Mitigation Training | Communication Training Only | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Customized [Count of Participants; unit: Participants]
  >18 years of age | 11 | 11 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 8 | 7 | 15
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22
Years in Practice [Count of Participants; unit: Participants] — The number of years in practice for physician providers enrolled into the study is summarized by study arm/group using ordinal variables.
  Participants
    Less than 5 years | 11 | 8 | 19
    5-10 years | 0 | 2 | 2
    Greater than 10 years | 0 | 1 | 1
Provider Specialty [Count of Participants; unit: Participants] — Provider specialty for physicians enrolled into the study is summarized by study arm/group using categorical variables.
  Participants
    Internist | 0 | 3 | 3
    Oncologist | 1 | 0 | 1
    Intensivist | 10 | 6 | 16
    Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Verbal Dominance
Description: Verbal dominance was determined by the ratio of clinician to caregiver speaking time during the encounter, ranging from a minimum of 0 to a maximum of approximately 3. A ratio of >1 indicates that the clinician dominated the discussion. Ratio of clinician to caregiver speaking times are expressed as decimals and summarized both prior to and following the intervention by study arm.
Time Frame: During the intervention, up to 5 hours
Population: One participant in the intervention arm withdrew due to time constraints.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Communication and Bias Mitigation Training | Communication Training Only
Number analyzed (Participants) | 11 | 11
ratio
  Pre-Intervention | 2.65 (0.95) | 2.57 (0.81)
  Post-Intervention: number analyzed (Participants) | 10 | 11
  Post-Intervention | 2.10 (0.88) | 1.74 (0.62)
Statistical Analysis 1: Comparison: Communication and Bias Mitigation Training vs Communication Training Only; Test type: Superiority; p = 0.34, t-test, 2 sided — t-test of the mean pre/post difference between study arms; Mean Difference (Net) = -0.47, 95% CI 2-sided [-1.48 to 0.53]; A 2-sided t-test of the mean pre/post difference between the two study arms was used

2. Secondary Outcome: Encounter Duration
Description: Encounter duration is an estimate of the time the physician speaks to the caregiver, ranging from 5 to 20 minutes, with higher scores indicating more engagement. Speaking time in minutes both prior to and following the intervention is summarized by study arm using basic descriptive statistics.
Time Frame: During the intervention, up to 5 hours
Population: One participant in the intervention arm withdrew due to time constraints.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Communication and Bias Mitigation Training | Communication Training Only
Number analyzed (Participants) | 11 | 11
minutes
  Pre-Intervention | 16.13 (2.55) | 17.55 (2.76)
  Post-Intervention: number analyzed (Participants) | 10 | 11
  Post-Intervention | 13.64 (3.73) | 16.00 (1.83)
Statistical Analysis 1: Comparison: Communication and Bias Mitigation Training vs Communication Training Only; Test type: Superiority; p = 0.27, t-test, 2 sided — t-test of mean pre/post difference between the 2 study arms; Mean Difference (Net) = 1.13, 95% CI 2-sided [-0.95 to 3.21]

3. Secondary Outcome: Verbal Communication
Description: Quality of verbal communication as rated by standardized (actor) caregiver using the three-item CollaboRATE tool which has a minimum score of 0 and maximum of 30 with higher scores indicating better communication. Scores prior to and following the intervention are summarized by study arm using basic descriptive statistics.
Time Frame: During the intervention, up to 5 hours
Population: One participant in the control arm withdrew due to time constraints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Communication and Bias Mitigation Training | Communication Training Only
Number analyzed (Participants) | 11 | 11
score on a scale
  Pre-Intervention | 7.5 (0.4) | 7.9 (0.7)
  Post-Intervention: number analyzed (Participants) | 10 | 11
  Post-Intervention | 6.0 (1.1) | 7.0 (0.7)
Statistical Analysis 1: Comparison: Communication and Bias Mitigation Training vs Communication Training Only; Test type: Superiority; p = 0.23, t-test, 2 sided — t-test of mean pre/post difference between study arms; Mean Difference (Net) = 1.55, 95% CI 2-sided [-1.08 to 4.18]

4. Secondary Outcome: Modified NAAS Score
Description: The Nonverbal Accommodation Analysis System is not a score, but rather a system of coding nonverbal communication behaviors, consisting of 10 behaviors, the results of which are individually reported below. We modified the system as planned in the proposed research by removing behaviors not found to be related to bias or to standardized caregiver outcomes. This resulted in removing the speech rate variable, but retaining the remaining 9 variables. We also modified the system to count all instances of each behavior during the entire encounter, rather than in 2-minute slices of time.
Time Frame: Duration of intervention, up to 5 hours
Population: Modified NAAS scores were not calculated instead individual components of the NAAS have been reported as separate outcome measures. This was done because the Nonverbal Accommodation Analysis System is not a score, but rather a system of coding nonverbal communication behaviors, consisting of 10 behaviors, the results for nine of which are individually reported below. There is no composite NAAS score in existence to calculate or report. The current protocol reflecting this has been uploaded.
Arm/Group | Communication and Bias Mitigation Training | Communication Training Only
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Physician Talk Time
Description: Physician talk time during the intervention was monitored and recorded. The mean duration of time the physician was speaking, both prior to and following the intervention, is summarized by study arm, adjusted by total duration of the encounter. The physician talk time is therefore given as a proportion of the total encounter duration and is expressed as a decimal unit.
Time Frame: During the intervention, up to 5 hours
Population: One participant in the intervention arm withdrew due to time constraints.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Communication and Bias Mitigation Training | Communication Training Only
Number analyzed (Participants) | 11 | 11
ratio
  Pre-Intervention | 0.65 (0.08) | 0.66 (0.06)
  Post-Intervention: number analyzed (Participants) | 10 | 11
  Post-Intervention | 0.55 (0.10) | 0.55 (0.08)
Statistical Analysis 1: Comparison: Communication and Bias Mitigation Training vs Communication Training Only; Test type: Superiority; p = 0.60, t-test, 2 sided — t-test of mean pre/post difference between study arms; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.09 to 0.06]

6. Secondary Outcome: Pauses
Description: Number of times per minute the participant paused their speech during the encounter, both prior to the and following the intervention, is summarized by study arm using basic descriptive statistics.
Time Frame: During the intervention, up to 5 hours
Population: One participant in the intervention arm withdrew due to time constraints.
Measure: Mean (Standard Deviation); unit: pauses per minute
Arm/Group | Communication and Bias Mitigation Training | Communication Training Only
Number analyzed (Participants) | 11 | 11
pauses per minute
  Pre-Intervention | 0.21 (0.18) | 0.25 (0.19)
  Post-Intervention: number analyzed (Participants) | 10 | 11
  Post-Intervention | 0.53 (0.30) | 0.38 (0.20)
Statistical Analysis 1: Comparison: Communication and Bias Mitigation Training vs Communication Training Only; Test type: Superiority; p = 0.24, t-test, 2 sided — t-test of the mean pre/post difference between study arms; Mean Difference (Net) = -0.18, 95% CI 2-sided [-0.49 to 0.13]

7. Secondary Outcome: Simultaneous Speech
Description: Number of times per minute that the subjects' speech overlapped with the standardized caregiver's speech, both prior to and following the intervention, is summarized by study arm using basic descriptive statistics.
Time Frame: During the intervention, up to 5 hours
Population: One participant in the intervention arm withdrew due to time constraints.
Measure: Mean (Standard Deviation); unit: instances of overlap per minute
Arm/Group | Communication and Bias Mitigation Training | Communication Training Only
Number analyzed (Participants) | 11 | 11
instances of overlap per minute
  Pre-Intervention | 0.21 (0.18) | 0.25 (0.19)
  Post-Intervention: number analyzed (Participants) | 10 | 11
  Post-Intervention | 0.53 (0.30) | 0.38 (0.20)
Statistical Analysis 1: Comparison: Communication and Bias Mitigation Training vs Communication Training Only; Test type: Superiority; p = 0.61, t-test, 2 sided — t-test of the mean pre/post difference between study arms; Mean Difference (Net) = 0.03, 95% CI 2-sided [-1.0 to 0.17]

8. Secondary Outcome: Number of Interruptions
Description: Number of times per minute the participant interrupted the standardized caregiver causing the standardized caregiver to stop speaking, both prior to and following the intervention, is summarized by study arm using basic descriptive statistics.
Time Frame: During the intervention, up to 5 hours
Population: One participant in the intervention arm withdrew due to time constraints.
Measure: Mean (Standard Deviation); unit: interruptions per minute
Arm/Group | Communication and Bias Mitigation Training | Communication Training Only
Number analyzed (Participants) | 11 | 11
interruptions per minute
  Pre-Intervention | 0.04 (0.08) | 0 (0)
  Post-Intervention: number analyzed (Participants) | 10 | 11
  Post-Intervention | 0.02 (0.04) | 0.04 (0.09)
Statistical Analysis 1: Comparison: Communication and Bias Mitigation Training vs Communication Training Only; t-test of the mean pre/post difference between study arms; Test type: Superiority; p = 0.11, t-test, 2 sided; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.02 to 0.15]

9. Secondary Outcome: Smiling
Description: Number of times per minute the participant smiled during the encounter, both prior to and following the intervention, is summarized by study arm using basic descriptive statistics.
Time Frame: During the intervention, up to 5 hours
Population: One participant in the intervention group left early due to time constraints and did not complete post-intervention measures.
Measure: Mean (Standard Deviation); unit: smiles per minute
Arm/Group | Communication and Bias Mitigation Training | Communication Training Only
Number analyzed (Participants) | 11 | 11
smiles per minute
  Pre-Intervention | 0.01 (0.02) | 0.15 (0.26)
  Post-Intervention: number analyzed (Participants) | 10 | 11
  Post-Intervention | 0.01 (0.02) | 0.09 (0.12)
Statistical Analysis 1: Comparison: Communication and Bias Mitigation Training vs Communication Training Only; t-test of mean pre/post difference between study arms; Test type: Superiority; p = 0.58, t-test, 2 sided; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.25 to 0.15]

10. Secondary Outcome: Laughing
Description: Number of times per minute the participant laughed during the encounter, both prior to and following the intervention, is summarized by study arm using basic descriptive statistics.
Time Frame: During the intervention, up to 5 hours
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: laughs per minute
Arm/Group | Communication and Bias Mitigation Training | Communication Training Only
Number analyzed (Participants) | 11 | 11
laughs per minute
  Pre-Intervention | 0 (0) | 0.02 (0.03)
  Post-Intervention: number analyzed (Participants) | 10 | 11
  Post-Intervention | 0.04 (0.08) | 0.04 (0.06)
Statistical Analysis 1: Comparison: Communication and Bias Mitigation Training vs Communication Training Only; t-test of mean pre/post difference between study arms; Test type: Superiority; p = 0.57, t-test, 2 sided; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.08 to 0.05]

11. Secondary Outcome: Gesturing
Description: Number of times per minute the participant gestured with their hands during the encounter, both prior to and following the intervention, is summarized by study arm using basic descriptive statistics.
Time Frame: During the intervention, up to 5 hours
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: gestures per minute
Arm/Group | Communication and Bias Mitigation Training | Communication Training Only
Number analyzed (Participants) | 11 | 11
gestures per minute
  Pre-Intervention | 3.87 (1.52) | 3.93 (1.85)
  Post-Intervention: number analyzed (Participants) | 10 | 11
  Post-Intervention | 2.84 (1.54) | 2.22 (1.41)
Statistical Analysis 1: Comparison: Communication and Bias Mitigation Training vs Communication Training Only; t-test of mean pre/post difference between study arms; Test type: Superiority; p = 0.76, t-test, 2 sided; Mean Difference (Net) = -0.24, 95% CI 2-sided [-1.87 to 1.38]

12. Secondary Outcome: Nodding
Description: Number of times per minute the participant nodded during the encounter, both prior to and following the intervention, is summarized by study arm using basic descriptive statistics.
Time Frame: During the intervention, up to 5 hours
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: nods per minute
Arm/Group | Communication and Bias Mitigation Training | Communication Training Only
Number analyzed (Participants) | 11 | 11
nods per minute
  Pre-Intervention | 2.68 (0.67) | 2.15 (0.78)
  Post-Intervention: number analyzed (Participants) | 10 | 11
  Post-Intervention | 2.53 (1.17) | 2.36 (1.36)
Statistical Analysis 1: Comparison: Communication and Bias Mitigation Training vs Communication Training Only; t-test of mean pre/post difference between study arms; Test type: Superiority; p = 0.29, t-test, 2 sided; Mean Difference (Net) = 0.48, 95% CI 2-sided [-0.44 to 1.42]

13. Secondary Outcome: Eye Contact
Description: This is a REVERSE CODED variable. It measures the proportion of time during the encounter that the participant was looking away from the standardized caregiver in seconds divided by total encounter time in seconds. Eye contact time, both prior to and following the intervention, is summarized by study arm using basic descriptive statistics.
Time Frame: During the intervention, up to 5 hours
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: proportion of time in seconds
Arm/Group | Communication and Bias Mitigation Training | Communication Training Only
Number analyzed (Participants) | 11 | 11
proportion of time in seconds
  Pre-Intervention | 0.005 (0.012) | 0.007 (0.012)
  Post-Intervention: number analyzed (Participants) | 10 | 11
  Post-Intervention | 0.014 (0.023) | 0.010 (0.024)
Statistical Analysis 1: Comparison: Communication and Bias Mitigation Training vs Communication Training Only; t-test of mean pre/post difference between arms; Test type: Superiority; p = 0.60, t-test, 2 sided; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.03 to 0.02]

ADVERSE EVENTS:
Time Frame: During the intervention, up to 5 hours.
Arm/Group | Communication and Bias Mitigation Training | Communication Training Only
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
This is a small pilot intervention that was underpowered to detect a meaningful difference in primary or secondary outcomes. The total duration of the encounter has limited informational value since many of the encounters were ended by the study team after a set amount of time due to time constraints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2026-01-20): https://cdn.clinicaltrials.gov/large-docs/88/NCT05165888/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-23): https://cdn.clinicaltrials.gov/large-docs/88/NCT05165888/ICF_001.pdf